CLINICAL TRIAL: NCT01393730
Title: Phase II Trial of Abiraterone Acetate Combined With Dutasteride With Correlative Assessment of Tumor Androgen Levels and Androgen Receptor Sequence and Signaling at Baseline and at Progression
Brief Title: Abiraterone Acetate Combined With Dutasteride for Metastatic Castrate Resistant Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mary-Ellen Taplin, MD (Other)
Responsible Party: Sponsor-Investigator, Mary-Ellen Taplin, MD, Associate Professor of Medicine, HMS, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-448
Record Dates: First submitted 2011-06-21; First posted 2011-07-13 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Prostate Cancer
Keywords: prostate; metastatic; castrate resistant
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Abiraterone Acetate; Dutasteride; Prednisone; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abiraterone+prednisone+dutasteride (Experimental): Abiraterone acetate 1000mg orally once per day + prednisone 5mg orally once per day for two months, followed by abiraterone 1000mg orally once per day + prednisone 5mg orally once per day + dutasteride 3.5mg orally once per day in 28-day cycles until symptomatic or radiographic progression
  Interventions: Drug: Abiraterone acetate; Drug: Dutasteride; Drug: Prednisone

INTERVENTIONS:
Drug: Abiraterone acetate
  Other Names: CB7630
Drug: Dutasteride
  Other Names: Avodart
Drug: Prednisone
  Other Names: Corticosteroid

SUMMARY:
The purpose of this research study is to determine if the addition of dutasteride to a regimen with abiraterone acetate and prednisone will improve on therapy in patients with castrate-resistant prostate cancer and metastatic disease. This study will also help determine the side effects of the study treatment and how often they occur.

DETAILED DESCRIPTION:
Patients will receive abiraterone acetate and prednisone orally, once daily for 2 months (2 cycles) on an outpatient basis. At the start of cycle 3, dutasteride will be taken once daily. Patients will return to the clinic on Day 14 of the first 3 cycles for routine blood tests.

Patients will come to the clinic every 12 weeks for a CT scan and/or x-ray of the chest, CT scan or MRI of the abdomen and pelvis, bone scan, and blood test for testosterone and other specialized blood test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of adenocarcinoma of the prostate
* Castrate resistant disease
* Metastatic disease
* Normal organ and marrow function
* Subjects with partners of childbearing potential must be willing to use adequate methods of birth control

Exclusion Criteria:

* Uncontrolled intercurrent illness
* Uncontrolled hypertension
* Active or symptomatic viral hepatitis or chronic liver disease
* History of pituitary or adrenal dysfunction
* Clinically significant heart disease
* History of a different malignancy unless disease-free for at least 5 years
* Known brain metastasis
* History of gastrointestinal disorders
* Prior therapy with abiraterone acetate
* HIV-positive individuals on antiretroviral therapy
* Requirement for steroid use greater than the equivalent of 5 mg of prednisone daily
* Atrial fibrillation or other cardiac arrhythmia requiring therapy
* Thromboembolism in the last 6 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-09; Primary Completion 2016-01 (Actual); Study Completion 2017-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, M.D., Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
This will not be done.

REFERENCES:
- [Result] McKay RR, Zukotynski KA, Werner L, Voznesensky O, Wu JS, Smith SE, Jiang Z, Melnick K, Yuan X, Kantoff PW, Montgomery B, Balk SP, Taplin ME. Imaging, procedural and clinical variables associated with tumor yield on bone biopsy in metastatic castration-resistant prostate cancer. Prostate Cancer Prostatic Dis. 2014 Dec;17(4):325-31. doi: 10.1038/pcan.2014.28. Epub 2014 Aug 5. PMID 25091040
- [Result] McKay RR, Werner L, Mostaghel EA, Lis R, Voznesensky O, Zhang Z, Marck BT, Matsumoto AM, Domachevsky L, Zukotynski KA, Bhasin M, Bubley GJ, Montgomery B, Kantoff PW, Balk SP, Taplin ME. A Phase II Trial of Abiraterone Combined with Dutasteride for Men with Metastatic Castration-Resistant Prostate Cancer. Clin Cancer Res. 2017 Feb 15;23(4):935-945. doi: 10.1158/1078-0432.CCR-16-0987. Epub 2016 Sep 28. PMID 27683182
- [Result] Chen EJ, Sowalsky AG, Gao S, Cai C, Voznesensky O, Schaefer R, Loda M, True LD, Ye H, Troncoso P, Lis RL, Kantoff PW, Montgomery RB, Nelson PS, Bubley GJ, Balk SP, Taplin ME. Abiraterone treatment in castration-resistant prostate cancer selects for progesterone responsive mutant androgen receptors. Clin Cancer Res. 2015 Mar 15;21(6):1273-80. doi: 10.1158/1078-0432.CCR-14-1220. Epub 2014 Oct 15. PMID 25320358
- [Derived] Wang Z, Deng T, Long X, Lin X, Wu S, Wang H, Ge R, Zhang Z, Wu CL, Taplin ME, Olumi AF. Methylation of SRD5A2 promoter predicts a better outcome for castration-resistant prostate cancer patients undergoing androgen deprivation therapy. PLoS One. 2020 Mar 5;15(3):e0229754. doi: 10.1371/journal.pone.0229754. eCollection 2020. PMID 32134978

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from September 2011 through October 2012
Groups:
- Abiraterone + Prednisone + Dutasteride: Abiraterone acetate + prednisone for two months, followed by abiraterone + prednisone + dutasteride in 28-day cycles until symptomatic or radiographic progression
  Abiraterone acetate: 1000 mg orally, once per day
  Dutasteride: 3.5 mg orally once per day
  Prednisone: 5 mg orally once per day
Period: Overall Study
Arm/Group | Abiraterone + Prednisone + Dutasteride
Started | 40
Treated | 38
Evaluable AR Amplification | 21
Evaluable AR Mutation | 14
Completed | 34
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Other | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [59 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Region of Enrollment [Number; unit: participants]
  United States | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Androgen Receptor (AR) Related Mutations
Description: AR related mutation was defined as presence of T878A mutation. Expression of T878A was measured by established methods.
Time Frame: Pairs of patients samples were evaluated at baseline and time of progression. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all patients evaluable for AR mutation.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 14
Participants | 1

2. Secondary Outcome: Change in Serum Levels of Testosterone
Description: Serum testosterone levels were estimated based on established methods. The change from baseline to progression was calculated for each participant.
Time Frame: Samples for testosterone analyses were obtained at baseline and at time of progression. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (Inter-Quartile Range); unit: ng/dL
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 38
ng/dL | 0.25 [0.1 to 0.5]

3. Secondary Outcome: Prostate-Specific Antigen (PSA) Response
Description: PSA response was defined as decline of 50% from baseline confirmed by a PSA at least 4 weeks later based on Prostate-specific Antigen Working Group-2 (PSAWG-2) (2008) criteria.
Time Frame: PSA was measured at baseline and day 1 of every cycle on treatment. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 38
Participants | 34

4. Secondary Outcome: Time to PSA Progression
Description: Time to PSA progression based on the Kaplan-Meier method was defined as the time between registration and documented PSA progression. PSA progression based on Prostate-Specific Antigen Working Group-2 (PSAWG-2) (2008) criteria was an increase of >/=25% and >/= 2 ng/ml after 12 weeks for patients without a PSA decline from baseline and an increase of >/=25% and >/= 2 ng/ml above the nadir, confirmed by a 2nd value 3 weeks or later for patients with a PSA decline from baseline. PSA progression was reported not duration of response.
Time Frame: as for outcome 3
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 38
months | 5 [3 to 8]

5. Secondary Outcome: Best Overall Response
Description: Overall response (OR) rate was defined as achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: Disease was evaluated radiologically at baseline and every 12 weeks cycles on treatment. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all treated patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 38
Participants | 6

6. Secondary Outcome: Time to Progression (TTP)
Description: TTP based on the Kaplan-Meier method is defined as the duration of time from study entry to documented first observation of progressive disease (PD). Per RECIST 1.0 for target lesions, PD is at least a 20% increase in sum LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or appearance of new lesions. For non-target lesions, PD is the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: Disease evaluation occurred every 12 weeks while patients were receiving treatment. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 38
Months | 11 [8 to 15]

7. Secondary Outcome: Presence of AR Amplification
Description: Presence of AR amplification was measured by established methods.
Time Frame: Patients' samples were evaluated at baseline and every 12 weeks on treatment. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all evaluable patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 21
Participants | 10

8. Secondary Outcome: Change in Serum Androgen Levels
Description: Serum androgen levels measured based on established methods. The change from baseline to progression was calculated for each participant.
Time Frame: Pairs of patients' samples for androgen analyses were obtained at baseline and at time of progression. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: The analysis dataset is comprised of all treated patients.
Measure: Median (Inter-Quartile Range); unit: ng/dl
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 38
ng/dl | 1.2 [0.7 to 2]

9. Secondary Outcome: Change in Circulating Tumor Cells (CTCs) Levels
Description: CTCs were measured based on established methods.
Time Frame: Pairs of patients' samples were evaluated at baseline and time of progression. In this study cohort, participants were followed up to 48 months for this endpoint.
Population: Data were not collected for this secondary endpoint.
Arm/Group | Abiraterone + Prednisone + Dutasteride
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. In this study cohort, participants were followed up to 48 months for this endpoint.
Description: Maximum grade toxicity by type for a patient over time including only treatment-related events (possible, probable or definite attribution) was first calculated. Patients appear once for a given toxicity type. Serious and Other Adverse Events (AEs) were defined as events of grades 3-5 and grades 1-2, respectively, based on Common Terminology Criteria for Adverse Events version 4 (CTCAEv4). 'Other' events have no further specification.
Arm/Group | Abiraterone + Prednisone + Dutasteride
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 12/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone + Prednisone + Dutasteride (N=38)
Alanine aminotransferase increased (Investigations) | 1
Lipase increased (Investigations) | 1
Conduction abnormality/Atrioventricular heart block - AV block-second degree Mobitz Type II (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Ureter (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Vagina (Infections and infestations) | 1
Thrombosis/embolism (vascular access-related) (Injury, poisoning and procedural complications) | 5
Thromboembolic event (Injury, poisoning and procedural complications) | 1
Lipase (Investigations) | 1
Bone: spine-scoliosis (Musculoskeletal and connective tissue disorders) | 2
"Neuropathy: cranial - CN III Pupil, upper eyelid, extra ocular movements" (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abiraterone + Prednisone + Dutasteride (N=38)
Bone marrow cellularity (Blood and lymphatic system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Blood/Bone Marrow-Other (Specify) (Blood and lymphatic system disorders) | 1
Conduction abnormality/Atrioventricular heart block - Wolff-Parkinson-White syndrome (Cardiac disorders) | 2
Palpitations (Cardiac disorders) | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1
External ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Ear and labyrinth disorders (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 2
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
"Fistula, GI - Anus" (Gastrointestinal disorders) | 1
"Fistula, GI - Esophagus" (Gastrointestinal disorders) | 7
"Fistula, GI - Ileum" (Gastrointestinal disorders) | 4
"Fistula, GI - Jejunum" (Gastrointestinal disorders) | 2
"Fistula, GI - Stomach" (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
"Obstruction, GI - Esophagus" (Gastrointestinal disorders) | 1
"Stricture/stenosis (including anastomotic), GI - Duodenum" (Gastrointestinal disorders) | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1
"Fatigue (asthenia, lethargy, malaise)" (General disorders) | 1
Obesity (General disorders) | 1
Sweating (diaphoresis) (General disorders) | 22
Weight gain (General disorders) | 3
Weight loss (General disorders) | 3
Localized edema (General disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Pain (General disorders) | 8
General disorders and administration site conditions - Other, specify (General disorders) | 1
Infection (documented clinically/microbiologically) w/Grade 3/4 neutrophils -Brain (Infections and infestations) | 2
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Liver (Infections and infestations) | 1
Infection (documented clinically or microbiologically) w/Grade 3 or 4 neutrophils -Nerve-peripheral (Infections and infestations) | 1
Infection (documented clinically or microbiologically) with Grade 3 or 4 neutrophils - Peristomal (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Infection (documented clinically/microbiologically) w/Grade 3/4 neutrophils -Upper aerodigestive NOS (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Bruising (Injury, poisoning and procedural complications) | 2
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 2
Fracture (Injury, poisoning and procedural complications) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 7
Alkaline phosphatase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 8
Blood bilirubin increased (Investigations) | 4
Anorexia (Metabolism and nutrition disorders) | 3
"Bicarbonate, serum-low" (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 1
"Glucose, serum-high (hyperglycemia)" (Metabolism and nutrition disorders) | 12
Bone: spine-scoliosis (Musculoskeletal and connective tissue disorders) | 3
Extremity-lower (gait/walking) (Musculoskeletal and connective tissue disorders) | 7
Extremity-upper (function) (Musculoskeletal and connective tissue disorders) | 5
Fibrosis-cosmesis (Musculoskeletal and connective tissue disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Local complication - device/prosthesis-related (Musculoskeletal and connective tissue disorders) | 2
"Muscle weakness, generalized or specific area (not due to neuropathy) - Extremity-upper" (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4
Soft tissue necrosis - Abdomen (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis - Head (Musculoskeletal and connective tissue disorders) | 1
Soft tissue necrosis - Neck (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal/Soft Tissue-Other (Specify) (Musculoskeletal and connective tissue disorders) | 2
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Irritability (children <3 years of age) (Nervous system disorders) | 1
"Leak, cerebrospinal fluid (CSF)" (Nervous system disorders) | 2
"Neuropathy: cranial - CN III Pupil, upper eyelid, extra ocular movements" (Nervous system disorders) | 2
Nervous system disorders (Nervous system disorders) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 4
Psychiatric disorders (Psychiatric disorders) | 1
"Leak (including anastomotic), GU - Kidney" (Renal and urinary disorders) | 4
"Leak (including anastomotic), GU - Spermatic cord" (Renal and urinary disorders) | 2
"Leak (including anastomotic), GU - Ureter" (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Gynecomastia (Reproductive system and breast disorders) | 2
Testicular pain (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Laryngeal fistula (Respiratory, thoracic and mediastinal disorders) | 1
Prolonged intubation after pulmonary resection (>24 hrs after surgery) (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2
Burn (Skin and subcutaneous tissue disorders) | 1
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Nail changes (Skin and subcutaneous tissue disorders) | 1
Rash: dermatitis associated with radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 1
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 3
Striae (Skin and subcutaneous tissue disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 4
Intra-operative injury - Pharynx (Surgical and medical procedures) | 1
Phlebitis (including superficial thrombosis) (Vascular disorders) | 2
Portal vein flow (Vascular disorders) | 10
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 15
Thrombosis/thrombus/embolism (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes